CLINICAL TRIAL: NCT05539391
Title: Effectiveness of an Optimisation Strategy for Emergency Tracheal Intubation on Postintubation Morbidity: A Cluster Randomized Controlled Trial
Brief Title: Optimisation Strategy for Emergency Tracheal Intubation
Acronym: OSETIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2021/25
Record Dates: First submitted 2022-08-04; First posted 2022-09-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Emergencies; Out-of-hospital Setting; Tracheal Intubation
Keywords: Out-of-hospital; Intubation; Complications; Vital distress; Rapid sequence intubation; Rocuronium; Gum Elastic Bougie
MeSH Terms: conditions — Emergencies | interventions — Restraint, Physical; Rapid Sequence Induction and Intubation; Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Combination rapid sequence intubation (RSI) with use of rocuronium and the bag-mask ventilation between induction and Gum Elastic Bougie GEB will be systematically used at the first attempt to facilitate intubation.
  Interventions: Other: Data patient; Other: Physical examination; Procedure: Rapid sequence intubation (RSI) : Rocuronium /Bag-mask ventilation /GEB
- Control Group (Active Comparator): Physicians will be reminded of the current recommendations for emergency intubation: Rapid sequence intubation (RSI) using succinylcholine and use of GEB to facilitate intubation in case of intubation failure under direct laryngoscopy.
  Interventions: Other: Data patient; Other: Physical examination; Procedure: Rapid sequence intubation (RSI) : Recommendations for emergency intubation

INTERVENTIONS:
Other: Data patient — Medical History and characteristic of patient
Other: Physical examination — Arterial pressure, arterial oxygen saturation, heart rate
Procedure: Rapid sequence intubation (RSI) : Rocuronium /Bag-mask ventilation /GEB — Rapid sequence intubation (RSI) will be performed with use of rocuronium as paralytic agent (1.2 mg/ kg). Bag-mask ventilation between induction and laryngoscopy will be performed. The GEB will be systematically used at the first attempt to facilitate intubation.
  Arms: Treatment group
Procedure: Rapid sequence intubation (RSI) : Recommendations for emergency intubation — Rapid sequence intubation (RSI) using succinylcholine as a paralytic agent (1 mg/kg), no systematic bag-mask ventilation between induction and laryngoscopy, use of GEB to facilitate intubation in case of intubation failure under direct laryngoscopy.
  Arms: Control Group

SUMMARY:
This study has to objective to assess, in adults' patients needing tracheal intubation because of vital distress, the effect of a combined strategy to reduce intubation-related morbidity. This strategy will associate systematic use of rocuronium as paralyzing agent to facilitate tracheal intubation, bag face-mask ventilation before intubation and Gum Elastic Bougie (GEB) use.

DETAILED DESCRIPTION:
Several studies have reported positive impact of some interventions on the tracheal intubation-related complications incidence. Providing bag face-mask ventilation between medication administration and initiation of laryngoscopy significantly reduced the number of peri intubation hypoxemia episodes. The use of a non-depolarizing (rocuronium) paralytic agent instead of succinylcholine is associated with less post-intubation complications occurrence. Finally, use of a tracheal tube introducer (GEB) as an aid for intubation in emergency patients with at least one prognostic factor of difficult laryngoscopy has been shown to facilitate intubation. Assessment of a strategy combining these three interventions to reduce intubation related morbidity in emergency situations has never been assessed. It is expected that the combination of these interventions will drastically reduce the morbidity associated with emergency intubation. The strategy assessed will associate rocuronium use as paralyzing agent to facilitate intubation, bag mask ventilation before intubation and GEB use at first intubation attempt in all patients. The emergency physician in charge of the patients will record out-of hospital outcomes immediately after the out-of-hospital period. Intra-hospital data will be retrieved from the patient's medical record on the 28th day after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient adult (≥ 18 years) presenting with vital distress requiring emergency tracheal intubation as assessed by the emergency physician in the out-of-hospital setting.
* Patient with all conditions (trauma, dyspnea, coma, overdoses, and shock) except those in cardiac arrest will be included.

Exclusion Criteria:

* Patient presenting of a contraindication to succinylcholine, and/or rocuronium, and/or sugammadex (rocunorium antagonist).
* Patient who have contraindication to bag face mask ventilation before intubation (ongoing emesis, hematemesis, or hemoptysis).
* Patient that are not members of a medical aid scheme (beneficiary or main member).
* Patient under specific protection measures: pregnant, parturient or nursing women; legal protection or deprived of liberty: patient under judicial protection, patient under guardianship/curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2023-01-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Severe intubation-related complications occurring during the first hour after intubation | Day 0
  Proportion of patients with severe intubation-related complications occurring during the first hour after intubation
  The severe intubation-related complications are:
  * Cardiac arrest.
  * At least one arterial hypotension episode defined by systolic blood pressure<90 mmHg.
  * At least one hypoxemia episode defined by an occurrence of a new episode of oxygen.
  * Saturation < 90%.
  * Severe cardiac arrhythmia: ventricular tachycardia.
  * Pulmonary aspiration, reported by the physician.
  * Esophageal intubation.
  * Unintentional extubation. Severe intubation-related complications will be recorded by the emergency physician in charge of the patient.

SECONDARY OUTCOMES:
Difficulty of the intubation process - Intubation Difficulty | Day 0
  Intubation Difficulty Score (IDS). minimum values is 0 and the maximum values is dependent on the added elements.
Difficulty of the intubation process - Intubation conditions assessed by the Copenhagen | Day 0
  Intubation conditions assessed by the Copenhagen score - The value is clinically not acceptable and clinical acceptable
Difficulty of the intubation process - Alternative techniques. | Day 0
  Proportion of patients intubated by alternative techniques.
Difficulty of the intubation process - Intubation attempts | Day 0
  Mean number of intubation attempts
Difficulty of the intubation process - Intubation failures under direct laryngoscopy. | Day 0
  Mean number of intubation failures under direct laryngoscopy.
Out-of hospital care -Time of out-of-hospital care | Day 0
  Mean time of out-of-hospital care (in minutes)
Out-of hospital care - sedative drugs | Day 0
  Mean total amount of sedative drugs used after intubation
Out-of hospital care - vasopressors | Day 0
  Mean total amount of vasopressors used after intubation
Out-of hospital care : Mortality | Day 0
  Out-of-hospital mortality.
Mortality | Day 28
  Vital status

CONTACTS AND LOCATIONS:
Overall Officials: Xavier COMBES, Pr, Principal Investigator — Université Hospital, Bordeaux
Locations (22):
- France (22):
  - CHU d'Angers, Angers
  - CH Carnelle Portes de l'Oise, Beaumont-sur-Oise
  - AP-HP - Hôpital Avicenne, Bobigny
  - CHU de Bordeaux - Hôpital Pellegrin, Bordeaux
  - CH de Pontoise René Dubos, Cergy-Pontoise
  - AP-HP - Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - GH Eaubonne Montmorency Hôpital Simone VEIL, Eaubonne
  - AP-HP - Hôpital Raymond Poincaré, Garches
  - CHU de Grenoble - Hôpital Nord La Tronche, La Tronche
  - CH de Versailles - Site André Mignot, Le Chesnay
  - HCL - Hôpital Edouard Herriot, Lyon
  - GH Sud Ile de France, Melun
  - CHU de Montpellier Site Lapeyronie, Montpellier
  - CHU de Nantes - Hôpital Hôtel Dieu, Nantes
  - AP-HP - Hôpital Lariboisière, Paris
  - AP-HP - Hôpital Pitié-Salpétrière, Paris
  - AP-HP - Hôpital Necker, Paris
  - CHU Poitiers - Hôpital la Milétrie, Poitiers
  - CHU de la Réunion - site Sud, Saint-Pierre
  - GH Sélestat Obernai, Sélestat
  - CHU Toulouse - Hôpital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No